CLINICAL TRIAL: NCT03143244
Title: Dexmedetomidine Versus Ketorolac/ Midazolam on Perioperative Outcome During Retinal Surgery.
Brief Title: Dexmedetomidine vs. Ketorolac/ Midazolam for Retinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS/15.12.26
Record Dates: First submitted 2017-04-15; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Retinal Surgery
MeSH Terms: interventions — Fumigant 93; Control Groups; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine group (D) (Active Comparator): Patients received 1ug/kg dexmedetomidine in 50 ml saline over 10 min i.v 30 min before induction then 0.4 ug/kg/h dexmedetomidine (4ug/ml) and normal saline 0.1 ml/kg till end of surgery, using two syringe pumps one for dexmedetomidine and the other for saline
  Interventions: Drug: Dexmedetomidine group (D)
- Ketorolac-Midazolam group (KM) (Active Comparator): Patients received 0.5mg/kg ketolac in 50 ml saline over 10 min before induction and 25ug/kg midazolam in 50 ml saline over 10 min i.v 30 min before induction then 50ug/kg/h of ketolac and 40ug/kg/h midazolam till end of surgery in two separate syringe pumps.
  Interventions: Drug: Ketorolac-Midazolam group (KM)
- Control group (Normal Saline) (C) (Placebo Comparator): Patients received same volume of normal slaine in two sets.
  Interventions: Drug: Control group (Normal Saline) (C)

INTERVENTIONS:
Drug: Dexmedetomidine group (D) — Patients received 1ug/kg dexmedetomidine in 50 ml saline over 10 min i.v 30 min before induction then 0.4 ug/kg/h dexmedetomidine (4ug/ml) and normal saline 0.1 ml/kg till end of surgery, using two syringe pumps one for dexmedetomidine and the other for saline
  Arms: Dexmedetomidine group (D)
Drug: Ketorolac-Midazolam group (KM) — Patients received 0.5mg/kg ketolac in 50 ml saline over 10 min before induction and 25ug/kg midazolam in 50 ml saline over 10 min i.v 30 min before induction then 50ug/kg/h of ketolac and 40ug/kg/h midazolam till end of surgery in two separate syringe pumps.
  Arms: Ketorolac-Midazolam group (KM)
Drug: Control group (Normal Saline) (C) — Patients received normal saline in two sets
  Arms: Control group (Normal Saline) (C)

SUMMARY:
To evaluate and compare the effect of administration of intravenous ketorolac- midazolam or dexmedetomidine as adjuvants to general anesthesia on perioperative outcome during retinal surgery.

DETAILED DESCRIPTION:
regarding patient registry; G power analysis was done was done to estimate the sample size. Assuming alpha (type I error) = 0.05 and beta (type II error) = 0.2 (power =80%), 18 patients per group would be sufficient to detect a difference 20 % in hemodynamics indices among the groups. A drop out 10% of cases was expected therefore 20 patients were required in each group to detect the difference.

- Statistical analysis: Data will be analyzed through SPSS (Statistical Package for Social Sciences). Program version 22. Distribution of data will be first tested by Kolmogorov-Smirnov test. Data is presented as mean and standard deviation (SD), median and range or numbers and percentages. For normally distributed data, one way ANOVA test will be used to compare between mean values of three groups with post hoc Bonferroni test for paired comparisons. Repeated measures ANOVA with post hock Bonferroni will be used for intra-groupal comparisons. For non-parametric data, Kruskal Wallis H test to compare between median values of 3 groups with Mann Whitney U test for paired comparisons. Chi Square test will be used for testing significance of categorical data. The P value ≤ 0.05 was considered as the level of statistical significance

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status |or ||

Exclusion Criteria:

* Mental disorders.
* Psychological disorders.
* Neurological disorders.
* Hyper reactive airway disease.
* History of sleep apnoea.
* Severe cardiovascular disease.
* Respiratory disease.
* Hepatic disease.
* Renal impairment.
* Known sensitivity to any of study drugs.
* History of alcohol.
* History of drug abuse.
* Morbid obesity (body mass index >35).
* Pregnancy.
* Lactating women.
* Patient refusal.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in blood pressure | for 8 hours after start of surgery
  Blood pressure measurements were performed electronically
Changes in heart rate | for 8 hours after start of surgery
  Heart rate measurements were performed electronically

SECONDARY OUTCOMES:
Intra-ocular pressure | for 8 hours after start of surgery
  Intra-ocular pressure was measured using tonometry technique
Occurrence of Oculao-cardiac reflex | for 14 hours after start of surgery
  Number of patients experienced intraoperative occulo-cardiac reflex
Postoperative nausea or vomiting | for 24 hours after start of surgery
  Number of patients experienced postoperative nausea or vomiting
Postoperative pain score | for 24 hours after start of surgery
  Numerical pain score ( for 24 hours after start of surgery) 0: non 1-3: mild 4-7: moderate 8-10: severe

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Abd el Motlb, MD, Study Director — Assisitant Professor

IPD SHARING:
Plan to Share IPD: Undecided